CLINICAL TRIAL: NCT06005948
Title: Investigation of the Effect of Dynamic Neuromuscular Stabilization on Pain, Functionality and Kinesiophobia in Individuals Undergoing Lumbar Disc Herniation Surgery
Brief Title: Investigation of the Effectiveness of Dynamic Neuromuscular Stabilization Exercises After Lumbar Disc Herniation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar75
Record Dates: First submitted 2023-08-15; First posted 2023-08-23 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain; Kinesiophobia
Keywords: pain; Neuromuscular Stabilization exercises; Kinesiophobia; surgical
MeSH Terms: conditions — Low Back Pain; Kinesiophobia; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The dynamic neuromuscular stabilization exercises
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): No exercise will be given after surgery
  Interventions: Other: control
- exercise group (Experimental): Dynamic neuromuscular stabilization exercises will be performed for 8 weeks after surgery.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — The dynamic neuromuscular stabilization group will receive developmental postures based on developmental kinesiology. It will involve a supine 3month Position, side-lying Position, Quadruped, oblique sitting, bear position, squat Position. Each position will be performed for 30-60 s for five reps, active exercise 5-10 reps under supervision for two days/week, and unsupervised for 3 days/week for 8 weeks
  Arms: exercise group
Other: control — No intervention will be made.
  Arms: control group

SUMMARY:
The aim of the study is to investigate the effects of dynamic neuromuscular stabilization exercises on pain, functionality and fear in individuals who have undergone lumbar disc herniation surgery.

DETAILED DESCRIPTION:
The research was planned as a randomized controlled trial, which is a quantitative study. Participants will be divided into 2 groups as control and exercise groups by simple randomization method. The individuals in the control group of the study will not be given any exercise program after surgery. A home exercise program created with Dynamic Neuromuscular Stabilization exercises after surgery will be applied to the individuals in the intervention group. Data collection will be carried out through an online survey. The scales and forms to be used before and after the treatment are respectively: 1. Oswestry Low Back Pain Disability Questionnaire 2. International Physical Activity Questionnaire (Short Form) 3. Questionnaire for Fear of Daily Living Activities The questionnaires will be uploaded to the Google Forms database and the participants will be accessed via e-mail or mobile phone applications. . They will be asked to fill out the questionnaires before starting the post-surgical exercise program and the exercise program will be explained practically before discharge. The exercises will be planned 3 times a week and for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be between 30 and 50 years old.
* Having undergone lumbar disc hernia surgery.
* Having access to a computer/tablet/phone and internet.

Exclusion Criteria:

* Having cognitive, mental or psychological problems.
* Having a visual or hearing impairment.
* Having a physical condition that causes significant loss of function

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
The Oswestry Disability Index | 10 weeks
  The questionnaire includes ten topics related to pain severity, weight lifting, self-care, walking, sitting, sexual function, standing, social life, sleep quality, and ability to travel. expression follows. The patient then checks for the expression that most closely resembles his condition. Each question is scored on a scale of 0-5, with the first statement being zero and indicating the least disability, and the last statement being scored as 5 indicating the most severe disability. The scores of all answered questions are added up, then multiplied by two to get the index (range 0 to 100). Zero equals no obstacle and 100 is the maximum possible obstacle.
International Physical Activity Questionnaire Short Form (IPAQ-SF) | 10 weeks
  It consists of 7 questions. The questions provide information about time spent walking, time spent in moderate and vigorous activities, and time spent sitting. Calculation of the short form's total score includes the sum of time (minutes) and frequency (days) of walking, moderate-intensity activity, and vigorous activity. The energy required for activities is calculated with the metabolic equivalent (MET) -minute score. Standard MET values have been established for these activities. These are; Sitting 1.5 MET, Walking 3.3 MET, Moderate-intensity physical activity 4.0 MET, Vigorous physical activity 8.0 MET. Daily and weekly physical activity using these values level is calculated.
Fear of Daily Living Activities Questionnaire | 10 weeks
  In the questionnaire consisting of 10 questions, the participant is asked to score each question between 0 and 100. No fear of the activity is set to 0 and excessive fear of the activity is 100. In addition, the participants are asked to add 2 different activities that are not included in the survey but cause fear.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra ARISÜT, Study Chair — Uskudar University
Locations (1):
- Uskudar university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venkatesan P, K S, Kishen TJ, Janardhan S, Kumar Cr S. Comparison of yoga and dynamic neuromuscular stabilization exercise in chronic low back pain on magnetic resonance imaging of lumbar multifidus- protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2022 May 28;28:100937. doi: 10.1016/j.conctc.2022.100937. eCollection 2022 Aug. PMID 35789639
- [Background] Baerga-Varela L, Abreu Ramos AM. Core strengthening exercises for low back pain. Bol Asoc Med P R. 2006 Jan-Mar;98(1):56-61. PMID 19610550
- [Background] Butowicz CM, Acasio JC, Silfies SP, Nussbaum MA, Hendershot BD. Chronic low back pain influences trunk neuromuscular control during unstable sitting among persons with lower-limb loss. Gait Posture. 2019 Oct;74:236-241. doi: 10.1016/j.gaitpost.2019.09.019. Epub 2019 Sep 18. PMID 31563825
- [Background] Kararti C, Ozsoy I, Ozyurt F, Basat HC, Ozsoy G, Ozudogru A. The effects of dynamic neuromuscular stabilization approach on clinical outcomes in older patients with chronic nonspecific low back pain: a randomized, controlled clinical trial. Somatosens Mot Res. 2023 Sep;40(3):116-125. doi: 10.1080/08990220.2023.2191705. Epub 2023 Mar 24. PMID 36964655
- [Background] Lariviere C, Gagnon DH, Henry SM, Preuss R, Dumas JP. The Effects of an 8-Week Stabilization Exercise Program on Lumbar Multifidus Muscle Thickness and Activation as Measured With Ultrasound Imaging in Patients With Low Back Pain: An Exploratory Study. PM R. 2018 May;10(5):483-493. doi: 10.1016/j.pmrj.2017.10.005. Epub 2017 Oct 31. PMID 29097271